CLINICAL TRIAL: NCT07068893
Title: A 4-Anchor Construct With Internal Bracing Technique for Surgical Treatment of Perilunate Dislocations: A Prospective Study
Brief Title: A 4-Anchor Construct With Internal Bracing Technique for Surgical Treatment of Perilunate Dislocations
Status: Recruiting | Type: Observational
Sponsor: Bryan D Brown,MD (Other)
Responsible Party: Sponsor-Investigator, Bryan D Brown,MD, Orthopedic Hand, Elbow & Shoulder Surgeon, Orlando Health, Inc.
Organization: Orlando Health, Inc. (Other)
Other Study IDs: 25.007.01
Record Dates: First submitted 2025-06-23; First posted 2025-07-16 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Perilunate Dislocation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who undergo traditional fixation
- Patients who undergo fixation using a novel 4-anchor construct with internal bracing

SUMMARY:
The purpose of the research study is to determine the overall clinical and radiographic outcome differences between internal brace technique and the gold standard Kirschner wires (K-wire) technique for treatment of perilunate dislocations (e.g. nonunion, reoperation, infection, fixation failure, etc.). A secondary purpose is to determine the specific types of complications and their incidence rates with respect to internal brace technique and the gold standard Kirschner wires (K-wire) technique (e.g. range of motion losses, pain, numbness, weakness, etc).

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients who have undergone surgical fixation of perilunate dislocation

Exclusion Criteria:

* Perilunate dislocations with concomitant carpal fracture(s)
* Pediatric patients (Age < 18 years-old)
* Patients whose age is greater than or equal to 89 years
* History of previous perilunate dislocation on ipsilateral side

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients, 18 years of age and older, who undergo operative fixation for perilunate dislocations without fracture at the level one trauma center, Orlando Health Orlando Regional Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Functional Assessment | From enrollment to 2-years postoperative
  assessment to measure wrist flexion/extension (degrees), wrist flexion/extension arc (degrees), and composite wrist function
Quick DASH Form | From enrollment to 2-years postoperative
  Assessment of symptoms and ability to perform certain activities.

SECONDARY OUTCOMES:
Specific types of complications and their incidence rates | From enrollment to 2-years postoperative
  Determine the specific types of complications and their incidence rates with respect to internal brace technique and the gold standard Kirschner wires (K-wire) technique (e.g. range of motion losses, pain, paresthesias, weakness, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided